CLINICAL TRIAL: NCT05737771
Title: A Phase 1 Clinical Trial to Compare and Evaluate the Safety and Pharmacokinetic Characteristics of the Fixed-dose Combination of DWJ1563 Compared to the Loose Combination of DWP16001 and DWC202213
Brief Title: To Compare the Pharmacokinetic Characteristics of the Fixed-dose Combination Compared to the Loose Combination
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWJ1563101
Record Dates: First submitted 2023-01-17; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: FDC; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Enavogliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Other): administrate DWP16001 + DWC202213 at first period, and administrate DWJ1563 at second period
  Interventions: Drug: DWC202213; Drug: DWJ1563; Drug: DWP16001
- Group B (Other): administrate DWJ1563 at first period, and administrate DWP16001 + DWC202213 at second period
  Interventions: Drug: DWC202213; Drug: DWJ1563; Drug: DWP16001

INTERVENTIONS:
Drug: DWC202213 — DWC202213
Drug: DWJ1563 — DWJ1563
Drug: DWP16001 — DWP16001

SUMMARY:
To compare the safety and pharmacokinetic properties between the administration of DWP16001 and DWC202213 as an individual drug, and the administration of DWJ1563 as a combination drug.

ELIGIBILITY:
Inclusion Criteria:

1. Before participating in the clinical trial, a person who fully explained the purpose, content, and characteristics of the clinical trial drug and signed a written consent form approved by the IRB of Chungbuk University Hospital to participate in this study according to his free will.
2. Healthy adults aged 19 or older at the time of screening.
3. Those who weigh more than 50.0 kg in men and women, and have a body mass index (BMI) of 18.0 kg/m2 or more and less than 30.0 kg/m2 or less in women.

   * Body mass index (BMI) = Weight (kg) / [Height (m)] 2.

Exclusion Criteria:

1. A person with a clinically significant history in liver, kidney, neuropsychiatric system, respiratory system, endocrine system, blood and tumor system, cardiovascular system (including orthostatic hypotension), digestive system, musculoskeletal system, etc.
2. A history of gastrointestinal diseases (e.g., esophageal diseases such as Crohn's disease, esophageal achalasia, or esophageal stenosis) or surgery (except appendectomy, hernia).
3. Those who are hypersensitive to other drugs (DPP-4 inhibitors, etc.) or have a history of clinically significant hypersensitivity reactions, including DWP16001, DWC202213 and homogeneous (SGLT2 inhibitors)
4. A person who shows the following results in the inspection items conducted during screening.

   * Blood ALT, AST, Total bilirubin > twice the upper limit of the normal range.
   * The glomerular filtration rate (e-GFR) <90 mL/min/1.73 m2 (using the CKD-EPI method)
5. After more than 3 minutes of rest, systolic blood pressure > 150 mmHg or <90 mmHg, or diastolic blood pressure > 100 mmHg or <60 mmHg, or pulse ≤ 40 bpm or ≥ 100 bpm in vital signs measured at the seat

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
AUC0-t of DWP16001 | 0 to 24 hours
  AUC0-t of DWP16001
Cmax of DWP16001 | 0 to 24 hours
  Cmax of DWP16001
AUC0-t of DWC202213 | 0 to 24 hours
  AUC0-t of DWC202213
Cmax of DWC202213 | 0 to 24 hours
  Cmax of DWC202213

CONTACTS AND LOCATIONS:
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, Seowon-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided